CLINICAL TRIAL: NCT03010839
Title: Cardiopulmonary Protection of Modified Remote Ischaemic Preconditioning in Mitral Valve Replacement Surgery
Brief Title: Cardiopulmonary Protective Effects of Modified Remote Ischaemic Preconditioning in Mitral Valve Replacement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Su Liu, M.D/Ph.D, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XYFY-2017-001
Record Dates: First submitted 2016-12-31; First posted 2017-01-05 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Myocardial Injury; Remote Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Remote Ischemic Preconditioning(mRIPC) (Active Comparator): modified RIPC was induced at 24 h, 12 h and 1 h before surgery to reinforce the protective effects of RIPC. The single RIPC protocol was induced by three cycles of upper-limb ischemia, a standard blood-pressure cuff was placed on the ringt upper arm, then inflated the cuff to 200 mm Hg for 5 minutes, followed by 5 min of cuff deflation.
  Interventions: Procedure: Modified Remote Ischemic Preconditioning
- Control (Placebo Comparator): Control group without remote ischemic preconditioning
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Modified Remote Ischemic Preconditioning — mRIPC will be induced at 24 h, 12 h and 1 h before surgery and once before induction of anesthesia by 3 cycles of 5-min upper limb ischemia and 5-min reperfusion using a blood-pressure cuff inflated to a pressure 200mmHg
  Other Names: mRIPC
  Arms: Modified Remote Ischemic Preconditioning(mRIPC)
Procedure: Control — Control group witnout remote ischemic preconditioning
  Arms: Control

SUMMARY:
During cardiac surgery with cardiopulmonary bypass , injury occurs to the heart muscle and the lung.The heart and lung injury is a serious complication ,which increases both mortality and morbidity of cardiac surgery .Remote ischemic preconditioning(RIPC) with transient upper limb ischemia/reperfusion is a novel, simple, cost-free,non-pharmacological and non-invasive strategy.Recent some trials suggested that RIPC could provide myocardial protection by reducing serum cardiac biomarkers,however, more recent multicenter studies[9-11] had failed to show the protective effects of RIPC with respect to the troponin release and lung injury.

Remote ischemic preconditioning (RIPC) is reported to have the early-phase and delayed-phase organ protective effects, whether the modified RIPC protocol induced repeatedly has the cardiopulmonary protective effect is still uncertain.

DETAILED DESCRIPTION:
modified RIPC was induced at 24 h, 12 h and 1 h before surgery to reinforce the protective effects of RIPC.The single RIPC protocol was induced by three cycles of upper-limb ischemia, a standard blood-pressure cuff was placed on the ringt upper arm, then inflated the cuff to 200 mm Hg for 5 minutes, followed by 5 min of cuff deflation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing heart surgery on cardiopulmonary bypass
2. Patients aged 18 years to 80 years

Exclusion Criteria:

1. Inability to give informed consent
2. Cardiogenic shock
3. Cardiac arrest on current admission
4. Left ventricular ejection fraction less than 30%
5. Current atrial fibrillation
6. Preoperative use of inotropics or mechanical assist device
7. Patients with significant hepatic dysfunction (Prothrombin>2.0 ratio)
8. Patients with known renal failure with a GFR<30 mL/min/1.73 m2
9. Patients with significant pulmonary disease (FEV1<40% predicted)
10. Recent myocardial infarction (within 7 days)
11. Recent systemic infection or sepsis (within 7 days)
12. Severe stroke (within 2 months)
13. Significant peripheral arterial disease affecting the upper limbs
14. Previous serious psychiatric disorders (e.g. schizophrenia, dementia)
15. Surgeries: cardiac transplantation, concomitant carotid endarterectomy , previous heart surgery,off-pump surgery, emergency surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-11-05 (Actual); Primary Completion 2018-01-10 (Actual); Study Completion 2018-03-10 (Actual)

PRIMARY OUTCOMES:
Troponin I serum release over 24 hours after surgery | 24 hours post surgery

SECONDARY OUTCOMES:
PaO2/FiO2 ratio over 24 hours after surgery | 24 hours post surgery
salveolar-arterial oxygen gradient over 24 hours after surgery | 24 hours post surgery
Inotrope score | 12 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Liu Su, M.D/Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available when this trial is finished and the article have been published.

REFERENCES:
- [Result] Domanski MJ, Mahaffey K, Hasselblad V, Brener SJ, Smith PK, Hillis G, Engoren M, Alexander JH, Levy JH, Chaitman BR, Broderick S, Mack MJ, Pieper KS, Farkouh ME. Association of myocardial enzyme elevation and survival following coronary artery bypass graft surgery. JAMA. 2011 Feb 9;305(6):585-91. doi: 10.1001/jama.2011.99. PMID 21304084
- [Result] JENNINGS RB, SOMMERS HM, SMYTH GA, FLACK HA, LINN H. Myocardial necrosis induced by temporary occlusion of a coronary artery in the dog. Arch Pathol. 1960 Jul;70:68-78. No abstract available. PMID 14407094
- [Result] Braunwald E, Kloner RA. Myocardial reperfusion: a double-edged sword? J Clin Invest. 1985 Nov;76(5):1713-9. doi: 10.1172/JCI112160. No abstract available. PMID 4056048
- [Result] Sullivan PJ, Sweeney KJ, Hirpara KM, Malone CB, Curtin W, Kerin MJ. Cyclical ischaemic preconditioning modulates the adaptive immune response in human limb ischaemia-reperfusion injury. Br J Surg. 2009 Apr;96(4):381-90. doi: 10.1002/bjs.6554. PMID 19283744
- [Result] Bolli R. The late phase of preconditioning. Circ Res. 2000 Nov 24;87(11):972-83. doi: 10.1161/01.res.87.11.972. PMID 11090541
- [Result] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Result] Przyklenk K, Bauer B, Ovize M, Kloner RA, Whittaker P. Regional ischemic 'preconditioning' protects remote virgin myocardium from subsequent sustained coronary occlusion. Circulation. 1993 Mar;87(3):893-9. doi: 10.1161/01.cir.87.3.893. PMID 7680290
- [Result] Gho BC, Schoemaker RG, van den Doel MA, Duncker DJ, Verdouw PD. Myocardial protection by brief ischemia in noncardiac tissue. Circulation. 1996 Nov 1;94(9):2193-200. doi: 10.1161/01.cir.94.9.2193. PMID 8901671
- [Result] Oxman T, Arad M, Klein R, Avazov N, Rabinowitz B. Limb ischemia preconditions the heart against reperfusion tachyarrhythmia. Am J Physiol. 1997 Oct;273(4):H1707-12. doi: 10.1152/ajpheart.1997.273.4.H1707. PMID 9362234
- [Result] Li G, Labruto F, Sirsjo A, Chen F, Vaage J, Valen G. Myocardial protection by remote preconditioning: the role of nuclear factor kappa-B p105 and inducible nitric oxide synthase. Eur J Cardiothorac Surg. 2004 Nov;26(5):968-73. doi: 10.1016/j.ejcts.2004.06.015. PMID 15519191
- [Result] Kharbanda RK, Mortensen UM, White PA, Kristiansen SB, Schmidt MR, Hoschtitzky JA, Vogel M, Sorensen K, Redington AN, MacAllister R. Transient limb ischemia induces remote ischemic preconditioning in vivo. Circulation. 2002 Dec 3;106(23):2881-3. doi: 10.1161/01.cir.0000043806.51912.9b. PMID 12460865
- [Result] Hausenloy DJ, Yellon DM. Remote ischaemic preconditioning: underlying mechanisms and clinical application. Cardiovasc Res. 2008 Aug 1;79(3):377-86. doi: 10.1093/cvr/cvn114. Epub 2008 May 2. PMID 18456674
- [Result] Sivaraman V, Pickard JM, Hausenloy DJ. Remote ischaemic conditioning: cardiac protection from afar. Anaesthesia. 2015 Jun;70(6):732-48. doi: 10.1111/anae.12973. Epub 2015 Feb 26. PMID 25961420
- [Result] Heusch G, Botker HE, Przyklenk K, Redington A, Yellon D. Remote ischemic conditioning. J Am Coll Cardiol. 2015 Jan 20;65(2):177-95. doi: 10.1016/j.jacc.2014.10.031. PMID 25593060
- [Result] Kerendi F, Kin H, Halkos ME, Jiang R, Zatta AJ, Zhao ZQ, Guyton RA, Vinten-Johansen J. Remote postconditioning. Brief renal ischemia and reperfusion applied before coronary artery reperfusion reduces myocardial infarct size via endogenous activation of adenosine receptors. Basic Res Cardiol. 2005 Sep;100(5):404-12. doi: 10.1007/s00395-005-0539-2. Epub 2005 Jun 17. PMID 15965583
- [Result] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Result] Venugopal V, Hausenloy DJ, Ludman A, Di Salvo C, Kolvekar S, Yap J, Lawrence D, Bognolo J, Yellon DM. Remote ischaemic preconditioning reduces myocardial injury in patients undergoing cardiac surgery with cold-blood cardioplegia: a randomised controlled trial. Heart. 2009 Oct;95(19):1567-71. doi: 10.1136/hrt.2008.155770. Epub 2009 Jun 8. PMID 19508973
- [Result] Thielmann M, Kottenberg E, Boengler K, Raffelsieper C, Neuhaeuser M, Peters J, Jakob H, Heusch G. Remote ischemic preconditioning reduces myocardial injury after coronary artery bypass surgery with crystalloid cardioplegic arrest. Basic Res Cardiol. 2010 Sep;105(5):657-64. doi: 10.1007/s00395-010-0104-5. Epub 2010 May 21. PMID 20495811
- [Result] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384
- [Result] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504
- [Result] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Result] Meybohm P, Bein B, Brosteanu O, Cremer J, Gruenewald M, Stoppe C, Coburn M, Schaelte G, Boning A, Niemann B, Roesner J, Kletzin F, Strouhal U, Reyher C, Laufenberg-Feldmann R, Ferner M, Brandes IF, Bauer M, Stehr SN, Kortgen A, Wittmann M, Baumgarten G, Meyer-Treschan T, Kienbaum P, Heringlake M, Schon J, Sander M, Treskatsch S, Smul T, Wolwender E, Schilling T, Fuernau G, Hasenclever D, Zacharowski K; RIPHeart Study Collaborators. A Multicenter Trial of Remote Ischemic Preconditioning for Heart Surgery. N Engl J Med. 2015 Oct 8;373(15):1397-407. doi: 10.1056/NEJMoa1413579. Epub 2015 Oct 5. PMID 26436208
- [Result] Hausenloy DJ, Candilio L, Evans R, Ariti C, Jenkins DP, Kolvekar S, Knight R, Kunst G, Laing C, Nicholas J, Pepper J, Robertson S, Xenou M, Clayton T, Yellon DM; ERICCA Trial Investigators. Remote Ischemic Preconditioning and Outcomes of Cardiac Surgery. N Engl J Med. 2015 Oct 8;373(15):1408-17. doi: 10.1056/NEJMoa1413534. Epub 2015 Oct 5. PMID 26436207
- [Result] Remote Preconditioning Trialists' Group; Healy DA, Khan WA, Wong CS, Moloney MC, Grace PA, Coffey JC, Dunne C, Walsh SR, Sadat U, Gaunt ME, Chen S, Tehrani S, Hausenloy DJ, Yellon DM, Kramer RS, Zimmerman RF, Lomivorotov VV, Shmyrev VA, Ponomarev DN, Rahman IA, Mascaro JG, Bonser RS, Jeon Y, Hong DM, Wagner R, Thielmann M, Heusch G, Zacharowski K, Meybohm P, Bein B, Tang TY. Remote preconditioning and major clinical complications following adult cardiovascular surgery: systematic review and meta-analysis. Int J Cardiol. 2014 Sep;176(1):20-31. doi: 10.1016/j.ijcard.2014.06.018. Epub 2014 Jun 27. PMID 25022819
- [Result] Lucchinetti E, Bestmann L, Feng J, Freidank H, Clanachan AS, Finegan BA, Zaugg M. Remote ischemic preconditioning applied during isoflurane inhalation provides no benefit to the myocardium of patients undergoing on-pump coronary artery bypass graft surgery: lack of synergy or evidence of antagonism in cardioprotection? Anesthesiology. 2012 Feb;116(2):296-310. doi: 10.1097/ALN.0b013e318242349a. PMID 22222469
- [Result] Hong DM, Lee EH, Kim HJ, Min JJ, Chin JH, Choi DK, Bahk JH, Sim JY, Choi IC, Jeon Y. Does remote ischaemic preconditioning with postconditioning improve clinical outcomes of patients undergoing cardiac surgery? Remote Ischaemic Preconditioning with Postconditioning Outcome Trial. Eur Heart J. 2014 Jan;35(3):176-83. doi: 10.1093/eurheartj/eht346. Epub 2013 Sep 7. PMID 24014392
- [Result] Johnsen J, Pryds K, Salman R, Lofgren B, Kristiansen SB, Botker HE. The remote ischemic preconditioning algorithm: effect of number of cycles, cycle duration and effector organ mass on efficacy of protection. Basic Res Cardiol. 2016 Mar;111(2):10. doi: 10.1007/s00395-016-0529-6. Epub 2016 Jan 14. PMID 26768477
- [Result] Yamaguchi T, Izumi Y, Nakamura Y, Yamazaki T, Shiota M, Sano S, Tanaka M, Osada-Oka M, Shimada K, Miura K, Yoshiyama M, Iwao H. Repeated remote ischemic conditioning attenuates left ventricular remodeling via exosome-mediated intercellular communication on chronic heart failure after myocardial infarction. Int J Cardiol. 2015 Jan 15;178:239-46. doi: 10.1016/j.ijcard.2014.10.144. Epub 2014 Oct 30. PMID 25464262